CLINICAL TRIAL: NCT07092540
Title: The Baby Duchenne Study: Characterizing Developmental and Clinical Outcomes in the First Three Years in Children With Duchenne Muscular Dystrophy
Acronym: BABY DUCHENNE
Status: Not yet recruiting | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Bo Hoon Lee, Assistant professor of neurology, University of Rochester
Other Study IDs: STUDY00009939; US Department of Defense (Other: US Army Medical Research Acquisition Activity)
Record Dates: First submitted 2025-07-22; First posted 2025-07-30 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
Keywords: New born screening
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Boys (0-3) of age diagnosed with DMD via new born screening

SUMMARY:
The aim of the BABY DUCHENNE study is to evaluate the natural history and characterize the early clinical outcomes in very young children (0-3 years) with Duchenne muscular dystrophy (DMD) identified by newborn screening programs.

ELIGIBILITY:
Inclusion Criteria:

* Male child between birth and 3.0 years of age at time of enrollment.
* A confirmed and documented pathogenic or likely pathogenic variant in the DMD gene following a positive newborn screen.
* Ability of parent/guardian to understand and provide written informed consent (signing Parental Permission and Consent Form).
* Willingness of parent/guardian to comply with the protocol Schedule of Activities, including all study site visits.

Exclusion Criteria:

* Female
* Presence of any confirmed genetic disease, other than DMD, that could impact early development, which, in the opinion of the PI, may confound interpretation of developmental progress.
* Presence of any significant medical condition (i.e., extreme prematurity, hypoxic ischemic encephalopathy) which, in the opinion of the PI, may confound interpretation of the clinical course of DMD.
* Inability/unwillingness of parent/guardian to provide written permission (sign PPF) or to comply with the protocol Schedule of Activities.

Ages: 0 Days to 3 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Study Population: Males with genetically confirmed diagnosis of DMD (Duchenne Muscular Dystrophy)
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Mean Change in Bayley Scales of Infant and Toddler Development, Fourth Edition (Bayley-4) Gross Motor Standard Score | Baseline to 36 months
  The Bayley Scales of Infant and Toddler Development, Fourth Edition (Bayley-4), Gross Motor domain measures age-appropriate motor abilities such as crawling, standing, and walking in children aged 1 to 42 months. The Gross Motor Standard Score is derived by converting raw scores to age-normed standard scores (mean = 100; standard deviation = 15). Higher scores indicate better gross motor development.

SECONDARY OUTCOMES:
Mean Change in Bayley Scales of Infant and Toddler Development, Fourth Edition (Bayley-4) Cognitive Standard Score | Baseline to 36 months
  The Bayley-4 Cognitive domain measures early cognitive development, including attention, memory, and problem-solving abilities. Standard scores range from 40 to 160 (mean = 100; standard deviation = 15). Higher scores reflect better cognitive performance.
Mean Change in Bayley Scales of Infant and Toddler Development, Fourth Edition (Bayley-4) Fine Motor Standard Score | Baseline to 36 months
  The Bayley-4 Fine Motor domain assesses hand and finger coordination tasks such as reaching and grasping. Standard scores range from 40 to 160 (mean = 100; standard deviation = 15). Higher scores indicate better fine motor development.
Mean Change in Bayley Scales of Infant and Toddler Development, Fourth Edition (Bayley-4) Expressive Language Standard Score | Baseline to 36 months
  The Bayley-4 Expressive Language Standard Score is derived by converting raw scores to age-normed standard scores based on normative data for children ages 1 to 42 months. Standard scores range from 40 to 160, with a mean of 100 and a standard deviation of 15. Higher scores indicate more advanced expressive language abilities.
Mean Change in Bayley Scales of Infant and Toddler Development, Fourth Edition (Bayley-4) Receptive Language Standard Score | Baseline to 36 months
  The Bayley-4 Receptive Language domain assesses a child's ability to understand spoken language. Scores range from 40 to 160 (mean = 100; SD = 15). Higher scores reflect better language comprehension.
Mean Change in World Health Organization Motor Milestone (WHOMM) Checklist Score | Baseline to 36 months
  The WHO Motor Milestone (WHOMM) checklist records developmental attainment of 6 gross motor milestones, scored as achieved or not achieved. The score reflects the number of milestones achieved at each visit. Higher scores indicate greater motor milestone attainment for age.
Percentage of Participants Receiving Early Intervention Services | Baseline to 36 months
  This outcome measures the proportion of participants who have initiated any early intervention service (e.g., physical, occupational, or speech therapy), based on caregiver report or medical record review.
Age at Initiation of Early Intervention Services | Baseline to 36 months
  This outcome records the age (in months) at which participants first received early intervention services, based on caregiver report or documentation in the medical record.
Percentage of Participants Initiating Duchenne Muscular Dystrophy-Targeted Pharmacologic Treatment | Baseline to 36 months
  This outcome measures the proportion of participants who began any DMD-targeted pharmacologic treatment (e.g., corticosteroids, exon-skipping therapies) during the study period, based on caregiver report or medical records.
Age at Initiation of Duchenne Muscular Dystrophy-Targeted Pharmacologic Treatment | Baseline to 36 months
  This outcome records the age (in months) at which each participant initiated pharmacologic treatment for Duchenne Muscular Dystrophy, as reported by caregivers or documented in the medical record.
Percentage of Participants With a Neurobehavioral Diagnosis | Baseline to 36 months
  This outcome reports the percentage of participants diagnosed with a neurobehavioral condition (e.g., autism spectrum disorder, ADHD) during the study, based on caregiver report or medical record review.
Age at First Neurobehavioral Diagnosis | Baseline to 36 months
  This outcome records the age (in months) at which each participant received their first neurobehavioral diagnosis, as determined by caregiver report or medical record.
Mean Change in Duchenne Muscular Dystrophy Caregiver Reported Health Index Short Form (DMD-HI-SF) Score | Baseline to 36 months
  The DMD Caregiver Reported Health Index Short Form (DMD-HI-SF) is a caregiver-reported questionnaire assessing burden related to the child's health. Total score is derived by summing item responses and converting to a standardized T-score. Higher scores indicate greater symptom burden.
Baseline North Star Ambulatory Assessment (NSAA) Total Score at Age 3 Years | Baseline to 36 months
  The NSAA is a 17-item clinician-rated motor function scale validated for ambulant children with DMD. Each item is scored from 0 (unable) to 2 (normal), for a total score range of 0 to 34. A single NSAA total score will be recorded at the time of the participant's first assessment at age 3 years.